CLINICAL TRIAL: NCT07267065
Title: An Open-label Safety and Efficacy Study of AAV2-hAADC Administered by MRI-Guided Convective Infusion Using a Transfrontal Trajectory Into the Putamen and Caudate of Participants With Young Onset Parkinson's Disease
Brief Title: AAV2-hAADC for Parkinson's Disease (PDCS-01)
Acronym: PDCS-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Krzysztof Bankiewicz (Other)
Responsible Party: Sponsor-Investigator, Krzysztof Bankiewicz, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20251920
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease (PD); Early Onset Parkinson Disease
Keywords: Gene Therapy; AAV2-hAADC
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: The current study is an open-label dose escalation study investigating the safety and efficacy of 2 dose levels of AAV2-hAADC in participants with PD and fluctuating responses to levodopa. Up to 9 participants are planned to be enrolled and treated on Day 0.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Low Dose) (Experimental): Total Dose (vg): up to 4.2E12
  Interventions: Drug: AAV2-hAADC
- Dose 2 (High Dose) (Experimental): Total Dose (vg): up to 1.3E13
  Interventions: Drug: AAV2-hAADC

INTERVENTIONS:
Drug: AAV2-hAADC — The purpose of this study is to investigate AAV2-hAADC gene therapy (the study drug) for the treatment of moderately-advanced PD with motor fluctuations.
  AAV2-hAADC gene therapy works by using a modified virus called adeno-associated virus 2 (AAV2). This virus is naturally-occurring and not associated with any disease. The virus' DNA has been changed so that it can deliver the human enzyme called Aromatic L-Amino Acid Decarboxylase (AADC). This enzyme converts levodopa into dopamine. AAV2-hAADC can enter brain cells and transfer the copy of the AADC gene directly into these cells. Once the gene is inside the brain cells, those cells will make AADC. By increasing the levels of AADC, we aim to increase the levels of dopamine and improve the symptoms of PD.
  AAV2-hAADC will be delivered through a brain surgery to two parts of the brain called the putamen and the caudate. These parts of the brain are involved in PD.
  The goal of this study is to assess whether infusing AAV2-h

SUMMARY:
This study is looking at whether a gene therapy called AAV2-hAADC is safe and may help people with Parkinson's Disease.

AAV2-hAADC is intended to increase the levels of dopamine in your brain. It contains a virus called adeno-associated virus 2 (AAV2) that has been modified to carry the genetic code for an enzyme called Aromatic L-Amino Acid Decarboxylase, or AADC for short.

In this study, AAV2-hAADC is delivered to two parts of the brain called the putamen and the caudate. Increasing the amount of AADC gene in these parts of the brain converts more levodopa into dopamine, the chemical that is lacking in PD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults 18-75 years of age (inclusive), at the time of signing the informed consent.
2. Diagnosed with idiopathic Parkinson's Disease as defined by the following:

   a. Presence of bradykinesia PLUS any of the following: i. Rigidity ii. Resting tremor iii. Postural instability
3. Disease duration since diagnosis of >3 years.
4. Patient reported symptom onset prior to the age of 50 (inclusive).
5. Modified Hoehn & Yahr Staging ≥2.5 in the practically defined OFF medication state (≥ 12 hours from last dose of anti-parkinsonian medications)
6. Disabling motor complications with an average of ≥3 hours of OFF time per day during waking hours within 7 days of the screening visit as confirmed by the Parkinson's Disease (PD) diary.
7. International Parkinson and Movement Disorder Society (MDS) Unified Parkinson's Disease Rating Scale (UPDRS) Part III (total motor) score ≥25 in the clinically defined OFF state.
8. Unequivocal responsiveness to dopaminergic therapy for a minimum of 1 year, including a 30% or greater improvement in the UPDRS III (motor score) between ON and OFF states, as determined by the Investigator after overnight withdrawal of Parkinson's medications.
9. In the judgment of the Investigator, a stable, optimal regimen of Parkinson's medications for at least 4 weeks prior to screening evaluation.
10. In the judgment of the Investigator, stable Parkinson's features and symptoms for at least 4 weeks prior to screening evaluation.
11. Laboratory values prior to surgery:

    1. Platelets >100E9/L (transfusion independent)
    2. Prothrombin time (PT)/partial thromboplastin time (PTT) in normal range and international normalized ratio (INR) ≤1.3
    3. Absolute neutrophil count >1.5E9/L
    4. Hemoglobin >10.0 g/dL
    5. Aspartate aminotransferase or alanine aminotransferase <2.5U/L × the upper limit of normal
    6. Total bilirubin <2.5 mg/dL
    7. Serum creatinine ≤1.5 mg/dL
    8. Hematocrit >34%
    9. White blood cell count <12E9/L
    10. Estimated glomerular filtration rate ≥30 mL/min.
12. Medically and cognitively capable of comprehending and signing the informed consent, as well as undergoing and complying with the surgical procedure and protocol requirements as determined by review of medical records, medical history, and clinical evaluation.
13. Ability to travel to study visits alone or able to designate a care partner who agrees to accompany the participant to study visits as determined by discussion with the participant, care partner (if applicable), and Investigator.
14. Agrees to defer any neurological surgery, including deep brain stimulation, until the 12-month study visit is completed.

Exclusion Criteria:

1. Atypical or secondary parkinsonism, including but not limited to symptoms resulting from trauma, brain tumor, infection, cerebrovascular disease, other neurological disease, or to drugs, chemicals, or toxins, as determined by the Investigator.
2. Presence of clinically significant cognitive impairment as defined by a Montreal Cognitive Assessment (MoCA) score of less than 241 at screening and/or clinical diagnosis of dementia by Investigator based on MoCA diagnostic criteria.
3. Presence or history of psychosis, except for minor psychosis.
4. Presence of severe depression, as indicated by a BDI-II score >28 within 5 years of screening evaluation.
5. Active suicidal ideation as indicated by positive response to items 4 or 5 on the screening C-SSRS, or any history of a suicide attempt
6. Presence of impulse control disorder, defined as a total score ≥10 on the Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS).
7. History of substance use disorder within 2 years of screening evaluation, as determined from interview with the participant and/or review of medical records.
8. Brain imaging abnormalities in the striatum or other regions that would substantially increase risk of surgery in the opinion of the investigator.
9. Contraindication to magnetic resonance imaging (MRI) and/or gadolinium (e.g., ProHance [gadoteridol]).
10. Coagulopathy or inability to temporarily stop any anticoagulation or antiplatelet therapy for at least 2 weeks during the perioperative period.
11. Prior stereotactic brain surgery including lesioning procedures, deep brain stimulation, infusion therapies or any other prior brain surgery that could complicate the study procedure and/or negatively impact study evaluations as determined from participant interview, screening MRI, and/or review of medical records.
12. Prior gene transfer, as determined from participant interview or review of medical records.
13. History of stroke, poorly controlled or significant cardiovascular disease, diabetes, or any other acute or chronic medical condition that would unreasonably increase the risks of the study procedures, as determined from interview with the participant and/or review of medical records.
14. History of malignancy other than treated carcinoma in situ within 3 years of screening evaluation.
15. Clinically apparent or laboratory-detected infection (including acute or chronic scalp infection) at the time of screening or baseline evaluations or immediately prior to surgery that would be a contraindication to surgery.
16. Prior or current treatment with any investigational agent within 5 half-lives or 30 days (whichever is shorter).
17. Any factors, medical or social, which would likely cause the inability to comply with the procedures of the protocol, including completion of Parkinson's Disease (PD) diaries, frequent and prolonged study visits (including off medication visits) and travel, in the judgment of the Investigator.
18. Chronic immunosuppressive therapy, including chronic steroids, immunotherapy, cytotoxic therapy, and chemotherapy as determined by participant interview and/or medical record.
19. Any serious medical condition or abnormal finding on physical examination or laboratory investigation that would substantially increase the risks of the study procedures in the opinion of the investigator.
20. Any medical condition that is likely to lead to disability during the study and interfere with or confound study assessments (including but not limited to orthopedic conditions, spinal disorders, neuropathy, myelopathy, severe pulmonary or cardiac disease, and compromised nutritional states), as determined from interview with the participant and/ or review of medical records.
21. Pregnant and lactating women.
22. Male or female with reproductive capacity who is unwilling to use barrier contraception for 6 months after surgery.
23. Ongoing treatments that might interfere with interpretation of the study outcome, including antipsychotic medications, apomorphine, or levodopa infusion therapy (Duopa).
24. Plans to participate in any other therapeutic intervention study within 12 months after surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Through 3 year Follow-up
  Assessment of AEs or SAEs and their relationship to the study procedure and study drug (graded as definite, probable, possible, unlikely, or unrelated).
MRI findings | Through Month 6 Follow-up
  Intraoperative and post-operative MRI findings
Physical Exam and labs | Through 3 year Follow-up
  Changes from baseline in physical examination findings and routine clinical laboratory analysis (hematology, clinical chemistries, immunologic assessments).
C-SSRS | Through 3 year Follow-up
  Changes in Columbia-Suicide Severity Rating Scale (C-SSRS) results

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No